CLINICAL TRIAL: NCT00893724
Title: The Effect of Supplemental Adjuvants for Intracellular Nutrition and Treatment on Diabetic Macular Edema and Neovascular Age-Related Macular Degeneration
Brief Title: Supplemental Adjuvants for Intracellular Nutrition and Treatment
Acronym: SAINTS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mid-Atlantic Retina Consultations, Inc. (Other)
Collaborators: West Virginia University (Other)
Responsible Party: Nabil M. Jabbour, MD, FACS/ Principal Investigator, Mid-Atlantic Retina Consultations, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FF0901
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema
Keywords: DME; NAMD; Oxidative damage; Nutritional supplements/vitamins; DNA repair; NAMD/wet AMD
MeSH Terms: interventions — Inosine; Tocopherols; Tocotrienols; Acetylcysteine; Niacinamide; Ascorbic Acid; Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- P (Placebo) (Placebo Comparator)
  Interventions: Drug: Neutral pills with no medicinal effect
- S (Supplement) (Active Comparator)
  Interventions: Dietary Supplement: Inosine; Tocopherols, Tocotrienol, CoQ10 combination capsule; Niacinamide SR; Viatmin C; N-acetyl Cysteine; Complete Multivitamin with all minerals
- SM (Supplement with Minocycline) (Active Comparator)
  Interventions: Drug: Inosine; Tocopherol, Tocotrienol, CoQ10 combination capsule; Niacinamide; Vitamin C; N-acetyl Cysteine; Complete Multivitamin with all minerals; Minocycline

INTERVENTIONS:
Drug: Neutral pills with no medicinal effect — Neutral pills with no medicinal effect
  Arms: P (Placebo)
Dietary Supplement: Inosine; Tocopherols, Tocotrienol, CoQ10 combination capsule; Niacinamide SR; Viatmin C; N-acetyl Cysteine; Complete Multivitamin with all minerals — Inosine [SR] - 1[500mg] tablet bid Tocopherols [200IU], Tocotrienol [10mg], CoQ10 [50mg] - combination capsule bid Sustained Release Niacinamide - 1 [750mg] tablet bid Vitamin C - 1 [1000mg] sustained release tablet bid N-acetyl Cysteine - 1 [600mg] sustained release tablet qd Complete Multivitamin with all minerals - 1 tablet (sustained release) bid
  Arms: S (Supplement)
Drug: Inosine; Tocopherol, Tocotrienol, CoQ10 combination capsule; Niacinamide; Vitamin C; N-acetyl Cysteine; Complete Multivitamin with all minerals; Minocycline — Inosine [SR] - 1 [500mg] tablet bid Tocopherol [200IU], Tocotrienol [10mg], CoQ10 [50mg] combination capsule bid Sustained Release Niacinamide 1 [750mg] tablet bid Vitamin C 1 [1000mg] sustained release tablet bid N-acetyl Cysteine 1 [600mg] sustained release tablet qd Complete Multivitamin with all minerals - 1 tablet (sustained release) bid Minocycline 1 [50mg] tablet qd
  Arms: SM (Supplement with Minocycline)

SUMMARY:
Nutritional supplements have an augmentative effect on the outcomes of standard treatment of diabetic macular edema (DME) and Neovascular Age-Related Macular Degeneration (NAMD).

DETAILED DESCRIPTION:
It has been shown that in chronic diseases, oxidative stress results from Nitric acid reacting with oxygen to form toxins that damage both somatic and mitochondrial DNA. The potential for protecting the DNA and promoting repair by using nutritional supplements will be tested by augmenting standard treatments for DME and NAMD with such supplements. The patients will be randomized to treatment group and placebo group and followed up for a year in a double masked fashion. Anatomic and visual outcomes, as well as side effects will be assessed and analyzed. If the results are promising, this pilot study can be used to design alternative (cheaper, better and longer lasting) treatments for DME, NAMD and perhaps other chronic illnesses.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of NAMD
* Clinical Diagnosis of DME

Exclusion Criteria:

* Pregnant Women
* Known allergy to any component used in the treatment combinations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-08 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Degree of regression (Optical Coherence Tomography) | Monthly
Duration of regression (Optical Coherence Tomography) | Monthly
Visual change (ETDRS) | Monthly

SECONDARY OUTCOMES:
Effect on HbA1C | Monthly
Effect on Blood pressure | Monthly
Effect on serum uric acid | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Jabbour, MD, FACS, Principal Investigator — M.A.R.C.
Locations (1):
- Mid-Atlantic Retina Consultations, Inc., Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300